CLINICAL TRIAL: NCT02690259
Title: Near Infrared Fluorescent Technique for Sentinel Lymph Node Mapping in Endometrial Cancer
Brief Title: Sentinel Lymph Node Detection in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RegionSkaneKKLund
Record Dates: First submitted 2015-11-05; First posted 2016-02-24 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Endometrial Neoplasms
Keywords: Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Detection of SLN followed by a complete lymphadenectomy. In this way every patients will serve as her own control
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentinel node procedure (Experimental): Enrolling all eligible endometrial cancer patient to the Sentinel node concept using indocyanine green.
  Interventions: Procedure: Sentinel node procedure

INTERVENTIONS:
Procedure: Sentinel node procedure — Patients with Endometrial cancer undergo Sentinel node procedure using Indocyanine green
  Other Names: Indocyanine green

SUMMARY:
In endometrial cancer (EC) pelvic and paraaortic lymphadenectomy is performed only in high risk groups (with approximately 20% of patients having lymph node metastases (LNM)) whereas no lymphadenectomy is recommended in low risk groups despite 5% LNM. Moreover, preoperative risk group allocation is known to be erroneous in up to 15% of patients.

A technique identifying sentinel lymph nodes (SLN) in endometrial cancer have the potential to spare extensive surgery in 80% of high risk patients, identify low risk patients with nodal metastases, diminish side effects caused by full lymphadenectomy and render some expensive preoperative risk group allocation measures unnecessary.

A clinically useful SLN technique requires a high technical success rate, a clear definition of SLN, an algorithm taking into account that metastatic nodes not always accumulate tracer and a reproducible surgical algorithm. A definition of SLN requires knowledge on lymphatic anatomy. Unfortunately all tracers, dyes/radiotracers often result in an abundance of colored/ signaling nodes. Therefore, a definition of a SLN requires identification of efferent/afferent lymph vessels.

Several publications describe sentinel node techniques in EC with a variety of tracers (various dyes, radiotracer, alone or in combination). Sentinel nodes are usually described as "radioactive nodes" or "colored nodes" only with no further discrimination. No study relate to an anatomical description of lymphatic pathways.

The aims of this study is to systematically display the major anatomical pathways with the use of ICG and to evaluate a standardized and reproducible SLN surgical algorithm based on lymphatic anatomy and identification of efferent lymph vessels.

DETAILED DESCRIPTION:
Endometrial cancer is an increasingly common gynecologic malignancy. The cumulative 5-year survival rate for node negative patients is 94%, 75% in those with metastatic pelvic lymph nodes only and 38% in patients with pelvic and paraaortic metastases. The proportion of node positive patients in adequately staged patient materials (usually high risk groups) is reported in the range of 15-21%. Depending on used risk criteria lymph node metastases occur in 1.5-7.8% in low risk patients. Some studies show better overall survival after pelvic and paraaortic lymphadenectomy, whereas other studies show increased complications with no survival benefit from the lymphadenectomy. Recent articles recommend paraaortic and pelvic lymp node metastases (LND) in high risk EC but the therapeutic value related to potential complications of nodal staging in EC is debated as well as how to define risk groups. An incidence of 0.9-5.2% severe lymphedema and 3.1% chylous ascites requiring treatment has been described after robotic pelvic and paraaortic lymphadenectomy.

The Sentinel node concept has been studied extensively in other cancer forms, for example breast and vulvar cancer. With the above mentioned controversy, patients with EC would benefit tremendously from a functioning Sentinel node concept. Studies using patent blue or radioactive tracer have not shown satisfactory results. The Da Vinci system (da Vinci® Surgical System, Intuitive Surgical Inc., Sunnyvale, Ca, USA) with Firefly technique could make a new concept possible in which major lymphatic drainage can be displayed and learned, hence allowing a standardization of SLN definitions. In our pilot studies, a reproducible surgical algorithm has been defined, overcoming and compensating the fact that ICG spreads quickly to several nodes.

Purpose: To develop a reliable Sentinel node Concept using the Firefly system with ICG in EC patients based on a defined lymphatic anatomy, a clear definition of a sentinel node and a reproducible surgical algorithm.

Hypothesis: The Firefly system using ICG enables the use of a Sentinel node concept in EC patients regardless risk group, so that only patients with pathologically proven lymph nodes metastases undergo a pelvic and paraaortic lymphadenectomy.

Methods of Research:

375 consecutive EC patients planned for robotic hysterectomy, bilateral salpingo-oophorectomy and in high risk patients also pelvic and paraaortic lymphadenectomy at Skane University Hospital, Lund, Sweden are enrolled in this study prospectively after giving written consent. The study is approved by the regional Institutional Review Board. With extended funding, the study will be expanded to another University Hospital in Sweden. Data on operative outcome, operative and postoperative complications, pathology reports and follow up for 24 months are prospectively collected. The use of Indocyanine green (ICG) and the Firefly system has the advantage of a fast uptake to lymphatic vessels and lymph nodes. Pilot studies have resulted in a new surgical method, standardization of operative technique and a clear definition of the Sentinel lymph node which now enables this study.

ELIGIBILITY:
Inclusion Criteria:

* Planned robotic operation due to endometrial carcinoma
* Patient suitable for laparoscopic surgery
* Signed consent

Exclusion Criteria:

* No consent
* Inability to understand study information
* surgical or anesthesiological contraindication for laparoscopic surgery
* previous lymphatic problems
* iodine allergy iodine
* disseminated disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Detection of sentinel nodes | up to 2 months
  The study measures the sensitivity of the described Sentinel node concept regarding the detection of Sentinel lymph nodes and detection of lymph node metastases
Detection of Sentinel nodes | up to 2 months
  The study measures the specificity of the described Sentinel node concept regarding the detection of Sentinel lymph nodes and detection of lymph node metastases
Detection of Setinel nodes | up to 2 months
  The study measures the false negative rate of the described Sentinel node concept regarding the detection of Sentinel lymph nodes and detection of lymph node metastases

SECONDARY OUTCOMES:
Recurrence rates | up to 24 months after inclusion
  The study measures the recurrence rate after concluded treatment including the Sentinel node concept
Lymphatic complications | up to 24 months after inclusion
  Comparison of the incidence of lymphatic complications such as lymph cysts and lymph edema after Sentinel node biopsy and full pelvic and paraaortic lymphadenectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Persson, Ass Prof, Study Director — Lund University
Locations (1):
- Department of Gynecology and Obstetrics, Lund, Sweden

REFERENCES:
- [Background] Geppert B, Persson J. Robotic infrarenal paraaortic and pelvic nodal staging for endometrial cancer: feasibility and lymphatic complications. Acta Obstet Gynecol Scand. 2015 Oct;94(10):1074-81. doi: 10.1111/aogs.12712. Epub 2015 Aug 25. PMID 26218968
- [Background] Schaafsma BE, van der Vorst JR, Gaarenstroom KN, Peters AA, Verbeek FP, de Kroon CD, Trimbos JB, van Poelgeest MI, Frangioni JV, van de Velde CJ, Vahrmeijer AL. Randomized comparison of near-infrared fluorescence lymphatic tracers for sentinel lymph node mapping of cervical cancer. Gynecol Oncol. 2012 Oct;127(1):126-30. doi: 10.1016/j.ygyno.2012.07.002. Epub 2012 Jul 10. PMID 22796548
- [Background] Holloway RW, Bravo RA, Rakowski JA, James JA, Jeppson CN, Ingersoll SB, Ahmad S. Detection of sentinel lymph nodes in patients with endometrial cancer undergoing robotic-assisted staging: a comparison of colorimetric and fluorescence imaging. Gynecol Oncol. 2012 Jul;126(1):25-9. doi: 10.1016/j.ygyno.2012.04.009. Epub 2012 Apr 13. PMID 22507531
- [Background] van der Vorst JR, Hutteman M, Gaarenstroom KN, Peters AA, Mieog JS, Schaafsma BE, Kuppen PJ, Frangioni JV, van de Velde CJ, Vahrmeijer AL. Optimization of near-infrared fluorescent sentinel lymph node mapping in cervical cancer patients. Int J Gynecol Cancer. 2011 Nov;21(8):1472-8. doi: 10.1097/IGC.0b013e31822b451d. PMID 22027751
- [Background] Rossi EC, Ivanova A, Boggess JF. Robotically assisted fluorescence-guided lymph node mapping with ICG for gynecologic malignancies: a feasibility study. Gynecol Oncol. 2012 Jan;124(1):78-82. doi: 10.1016/j.ygyno.2011.09.025. Epub 2011 Oct 11. PMID 21996262
- [Background] Rossi EC, Jackson A, Ivanova A, Boggess JF. Detection of sentinel nodes for endometrial cancer with robotic assisted fluorescence imaging: cervical versus hysteroscopic injection. Int J Gynecol Cancer. 2013 Nov;23(9):1704-11. doi: 10.1097/IGC.0b013e3182a616f6. PMID 24177256
- [Background] Jewell EL, Huang JJ, Abu-Rustum NR, Gardner GJ, Brown CL, Sonoda Y, Barakat RR, Levine DA, Leitao MM Jr. Detection of sentinel lymph nodes in minimally invasive surgery using indocyanine green and near-infrared fluorescence imaging for uterine and cervical malignancies. Gynecol Oncol. 2014 May;133(2):274-7. doi: 10.1016/j.ygyno.2014.02.028. Epub 2014 Feb 28. PMID 24582865
- [Background] How J, Gotlieb WH, Press JZ, Abitbol J, Pelmus M, Ferenczy A, Probst S, Gotlieb R, Brin S, Lau S. Comparing indocyanine green, technetium, and blue dye for sentinel lymph node mapping in endometrial cancer. Gynecol Oncol. 2015 Jun;137(3):436-42. doi: 10.1016/j.ygyno.2015.04.004. Epub 2015 Apr 12. PMID 25870917
- [Background] Plante M, Touhami O, Trinh XB, Renaud MC, Sebastianelli A, Grondin K, Gregoire J. Sentinel node mapping with indocyanine green and endoscopic near-infrared fluorescence imaging in endometrial cancer. A pilot study and review of the literature. Gynecol Oncol. 2015 Jun;137(3):443-7. doi: 10.1016/j.ygyno.2015.03.004. Epub 2015 Mar 11. PMID 25771495
- [Background] Sinno AK, Fader AN, Roche KL, Giuntoli RL 2nd, Tanner EJ. A comparison of colorimetric versus fluorometric sentinel lymph node mapping during robotic surgery for endometrial cancer. Gynecol Oncol. 2014 Aug;134(2):281-6. doi: 10.1016/j.ygyno.2014.05.022. Epub 2014 Jun 2. PMID 24882555
- [Derived] Luhrs O, Ekdahl L, Geppert B, Lonnerfors C, Persson J. Resection of the upper paracervical lymphovascular tissue should be an integral part of a pelvic sentinel lymph node algorithm in early stage cervical cancer. Gynecol Oncol. 2021 Nov;163(2):289-293. doi: 10.1016/j.ygyno.2021.08.031. Epub 2021 Sep 9. PMID 34509298
- [Derived] Luhrs O, Ekdahl L, Lonnerfors C, Geppert B, Persson J. Combining Indocyanine Green and Tc99-nanocolloid does not increase the detection rate of sentinel lymph nodes in early stage cervical cancer compared to Indocyanine Green alone. Gynecol Oncol. 2020 Feb;156(2):335-340. doi: 10.1016/j.ygyno.2019.11.026. Epub 2019 Nov 26. PMID 31780237

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02690259/Prot_SAP_000.pdf